CLINICAL TRIAL: NCT02651948
Title: Transperineal, MRI-guided, Prostate Biopsy: First Step to Focal Treatment of Prostate Cancer
Brief Title: Transperineal, MRI-guided, Prostate Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6253
Record Dates: First submitted 2015-12-23; First posted 2016-01-11 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transperineal prostate biopsy (TPB) (Experimental): Transperineal prostate biopsy MRI-guided
  Interventions: Procedure: Transrectal prostate biopsy (TRB):
- Transrectal prostate biopsy (TRB) (Active Comparator): Transrectal prostate biopsy echo-guided
  Interventions: Procedure: Transperineal, MRI-guided, prostate biopsy

INTERVENTIONS:
Procedure: Transperineal, MRI-guided, prostate biopsy
  Arms: Transrectal prostate biopsy (TRB)
Procedure: Transrectal prostate biopsy (TRB):
  Arms: Transperineal prostate biopsy (TPB)

SUMMARY:
Primary purpose:

Complications and rehospitalizations after transperineal prostate biopsy MRI-guided are reduced than transrectal prostate biopsies.

Secondary purposes:

* Patients tolerance after transperineal prostate biopsy MRI-guided is better than after transrectal prostate biopsies.
* Core of transperineal prostate biopsies are better than core of transrectal prostate biopsies
* Study of correlation between radiologic images and anatomopathologic result
* Description of needle track during the procedure
* Description of real time template saturation prostate biopsy
* Comparison of transperineal prostate biopsy relevance according to EBM
* Comparison of 1.5T MRI and 3T MRI for prostate cancer detection

ELIGIBILITY:
Inclusion criteria:

* Men
* 40 to 80 years' old
* Affiliation to French social health system
* Signed consent
* Prostate cancer suspicion based on prostate specific antigen (PSA) or digital rectal exam WITH abnormal MRI (Prostate Imaging Reporting and Data System score 3) AND negative transrectal prostate biopsies
* Patient treated by active surveillance for a low risk prostate cancer (T1c or T2a, Gleason = 6, PSA < 10)

Exclusion criteria:

* Gleason > 6 prostate cancer
* Metastatic prostate cancer
* Contraindication to MRI
* Contraindication to general anesthesia
* Non-reversible hemostasis trouble
* Inability to give consent

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Collection of complications and rehospitalizations by using questionnaire | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'urologie, Strasbourg, France

REFERENCES:
- [Result] Tricard T, Cazzato RL, Poussot B, Gaillard V, Labani A, De Mathelin M, Barhoumi C, Sauleau E, Gangi A, Roy C, Lang H. Transperineal MR Imaging-Guided Prostate Biopsy: A Prospective Randomized Controlled Study on Safety and Effectiveness Compared with Transrectal Biopsy. J Vasc Interv Radiol. 2025 Aug;36(8):1278-1284. doi: 10.1016/j.jvir.2025.05.015. Epub 2025 May 17. PMID 40389061